CLINICAL TRIAL: NCT06374628
Title: Pre-pectoral Tissue Expander and Acellular Dermal Matrix for a Two-stage Muscle Sparing Breast Reconstruction: Indications, Surgical Technique and Clinical Outcomes With Histological and Ultrasound Follow-up
Brief Title: Pre-pectoral Tissue Expander and Acellular Dermal Matrix for a Two-stage Muscle Sparing Breast Reconstruction
Status: Recruiting | Type: Observational
Sponsor: Rossella Elia, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Rossella Elia, MD PhD, Full time researcher, Unit of Plastic and Reconstructive Surgery, Policlinico of Bari, University of Bari
Organization: University of Bari (Other)
Other Study IDs: 0001
Record Dates: First submitted 2024-04-04; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: breast reconstruction — breast reconstruction in two-stages using tissue expander entirely wrapped by acellular dermal matrix

SUMMARY:
The aim of the research is to evaluate clinical outcomes of a two stage muscle sparing prepectoral breast reconstruction using tissue expander (TE) entirely covered by an ADM. The authors aim to report surgical indications, technical tips, clinical and histological outcomes with the final objective of delineate a decision-making algorithm for immediate prosthetic breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral mastectomy followed by two stage breast reconstruction with subcutaneous tissue expander and Acellular Dermal Matrix (ADM)
* risk-reducing mastectomies followed by two stage breast reconstruction with subcutaneous tissue expander and ADM

Exclusion Criteria:

* partial or total submuscular tissue expander placement,
* tissue expander placement in conjunction with latissimus dorsi muscle flap or without ADM, -delayed reconstructions
* previous breast surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients who undergo two stage breast recontrustion with tissue expander and ADM
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 24 months of follow-up
  Patients satisfaction will be evaluated through BREAST-Q questionnaire. the results from the questionnaire will be converted into a 0-100 scale with higher values meaning a better outcome

SECONDARY OUTCOMES:
Pain Evaluation | 24 months of follow-up
  Pain will be assessed trough Visual Analogic Scale (from minimum 0 to maximum 10). Higher values mean worse outcome

OTHER OUTCOMES:
Complication rate | 24 months of follow-up
  Complication will be recorded and classified with Clavien-Dindo Classification

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giudice, Study Director — University of Bari
Locations (1):
- AOU Policlinico, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided